CLINICAL TRIAL: NCT03563794
Title: Efficacy and Safety of Vildagliptin Added to Continuous Subcutaneous Insulin Infusion in Uncontrolled Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSII vs CSII+DPP-4 inhibitor
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: T2DM

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSII(insulin Lispro)+Vildagliptin (Experimental): Vildagliptin(50mg b.i.d po.) will be added to Continuous Subcutaneous Insulin Infusion(insulin Lispro) treatment in T2DM. Doses of insulin Lispro will be instructed on a titration schedule, adjusted every 2 days.
  Interventions: Drug: CSII+Vildagliptin
- CSII(insulin Lispro) (Active Comparator): T2DM patients will receive Continuous Subcutaneous Insulin Infusion(insulin Lispro) treatment. Doses of insulin Lispro will be instructed on a titration schedule, adjusted every 2 days.
  Interventions: Drug: CSII(insulin Lispro)

INTERVENTIONS:
Drug: CSII+Vildagliptin — Vildagliptin(50mg b.i.d po.) will be added to Continuous Subcutaneous Insulin Infusion(insulin Lispro) treatment in T2DM. Doses of insulin Lispro will be instructed on a titration schedule, adjusted every 2 days.
  Arms: CSII(insulin Lispro)+Vildagliptin
Drug: CSII(insulin Lispro) — T2DM patients will receive Continuous Subcutaneous Insulin Infusion(insulin Lispro) treatment. Doses of insulin Lispro will be instructed on a titration schedule, adjusted every 2 days.
  Arms: CSII(insulin Lispro)

SUMMARY:
The randomized, controlled clinical trial investigate the efficacy and safety of vildagliptin added to continuous subcutaneous insulin infusion in uncontrolled type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* T2DM
* 30≤ age≤70 years old
* BMI 18.0-28.0 Kg/m2
* HbA1c ≥8.5%
* Negtive GAD、ICA、IAA
* Patients do not use antihyperglycemia drugs
* Patients use antihyperglycemia drugs for ≥8 weeks(exclusion of DPP-4 inhibitors and GLP-1 receptor agonist)

Exclusion Criteria:

* T1DM,GDM
* Congestive heart failure (New York Heart Association Functional Classification III-IV)
* ALT or AST> 2 times above normal,GFR <50ml/min
* Severe infection in the previous 3 months
* Severely acute or chronic diabetic complications
* Patients who were taking medications,known to affect glycaemic control, such as glucocorticoids(aside from antidiabetic medications)
* History of pancreatitis
* Trauma or patients operating at a scheduled time
* Any mental health condition

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-06-10 (Estimated); Primary Completion 2019-06-10 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
blood glucose | 7 days
  changes from baseline in FPG and 2hPBG

SECONDARY OUTCOMES:
hypoglycemia | 7 days
  frequancy of hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- The first afilliated hospital of Xiamen university, Xiamen, Fujian, China